CLINICAL TRIAL: NCT01549587
Title: A Randomized Controlled Clinical Trial to Evaluate Late First to Mid-Second Trimester Introduction of Advanced Daily Oral Hygiene on Gingivitis and Maternity Outcomes
Brief Title: Oral Hygiene and Maternity Outcomes Multicenter Study (OHMOM)
Acronym: OHMOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011001
Record Dates: First submitted 2012-02-28; First posted 2012-03-09 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Gingivitis; Pregnancy
MeSH Terms: conditions — Gingivitis | interventions — Sodium Fluoride; Dental Devices, Home Care; Tin Fluorides; Cetylpyridinium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regular Oral Hygiene (Active Comparator): toothpaste, toothbrush and dental floss
  Interventions: Drug: 0.243% sodium fluoride; Device: toothbrush; Device: dental floss
- Advanced Oral Hygiene plus counseling (Experimental): toothpaste, toothbrush, mouth rinse and dental floss plus specialized education
  Interventions: Drug: 0.454% stannous fluoride; Device: toothbrush; Drug: 0.07% Cetylpyridinium chloride; Device: dental floss

INTERVENTIONS:
Drug: 0.243% sodium fluoride — dentifrice: brush thoroughly twice daily
  Other Names: Crest® Cavity Protection toothpaste
  Arms: Regular Oral Hygiene
Device: toothbrush — brush thoroughly twice daily
  Other Names: Oral-B® Indicator toothbrush, regular, soft
  Arms: Regular Oral Hygiene
Device: dental floss — floss the whole mouth once daily
  Other Names: Oral-B® Essentials dental floss
  Arms: Regular Oral Hygiene
Drug: 0.454% stannous fluoride — dentifrice: twice daily brush thoroughly for 2 minutes
  Other Names: Crest® Pro-Health toothpaste
  Arms: Advanced Oral Hygiene plus counseling
Device: toothbrush — twice daily brush thoroughly for 2 minutes
  Other Names: Oral-B® ProfessionalCare Series 1000 toothbrush, Oral-B® Precision Clean brush head
  Arms: Advanced Oral Hygiene plus counseling
Drug: 0.07% Cetylpyridinium chloride — mouth rinse: rinse with 20 mL of mouth rinse for 30 seconds twice daily
  Other Names: Crest® Pro-Health Multi-Protection Mouth Rinse
  Arms: Advanced Oral Hygiene plus counseling
Device: dental floss — floss the whole mouth once daily
  Other Names: Glide® Pro-Health Deep Clean dental floss
  Arms: Advanced Oral Hygiene plus counseling

SUMMARY:
This study will track changes in oral health in pregnant women. Subjects will be assigned to either regular oral care or advanced oral care and be given oral care products to use until they deliver. A comparison between the two groups (regular and advanced oral care) will be made to see if the oral care products impacted oral health and maternity variables.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* be at least the age of legal consent;
* be between 8 and 24 weeks of pregnancy;
* have at least 20 natural teeth;
* have moderate-to-severe gingivitis during pregnancy, including at least 30 intraoral sites with evidence of marginal gingival bleeding.

Exclusion Criteria:

* evidence of multiple gestations;
* history of HIV infection, AIDS, autoimmune disease, or diabetes other than gestational diabetes;
* indication for use of antibiotic pre-medication prior to dental procedures;
* systemic corticosteroid or immunosuppressive therapy within 1 month of Baseline;
* severe periodontal disease, rampant untreated dental caries, or other oral conditions that necessitate immediate dental care;
* ongoing dental care that in the opinion of the investigator could impact study participation;
* a history of allergies or hypersensitivity to mouth rinse products containing CPC;
* any disease or condition that in the opinion of the investigator could interfere with the safe completion of the study;
* randomization to a treatment in study 2011001 during a prior pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Jeffcoat, DMD, Principal Investigator — School of Dentistry University of Pennsylvania; Michael Reddy, DMD, DMSc, Principal Investigator — School of Dentistry University of Alabama
Locations (2):
- United States (2):
  - Center for Women's Reproductive Health, Birmingham, Alabama
  - Penn OB/Gyn and Associates, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Parry S, Jeffcoat M, Reddy MS, Doyle MJ, Grender JM, Gerlach RW, Tanna N, Geisinger ML, Geurs NC, Biggio J. Evaluation of an advanced oral hygiene regimen on maternity outcomes in a randomized multicenter clinical trial (Oral Hygiene and Maternity Outcomes Multicenter Study). Am J Obstet Gynecol MFM. 2023 Aug;5(8):100995. doi: 10.1016/j.ajogmf.2023.100995. Epub 2023 Apr 29. PMID 37127210

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Started | 373 | 373
Completed | 334 | 336
Not Completed | 39 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling | Total
Number analyzed (Participants) | 373 | 373 | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.6 (5.89) | 27.4 (6.01) | 27.46 (5.945)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 373 | 373 | 746
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 2 | 0 | 2
  Asian Oriential | 8 | 15 | 23
  Black | 260 | 262 | 522
  Caucasian | 76 | 77 | 153
  Hispanic | 13 | 10 | 23
  Asian Indian | 6 | 4 | 10
  Multi-racial | 8 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Löe-Silness Gingivitis Index
Description: Score Criteria 0 Normal gingiva.
  1. Mild inflammation - slight change in color, slight edema. No bleeding on probing.
  2. Moderate inflammation - redness, edema, and glazing. Bleeding on probing.
  3. Severe inflammation - marked redness, edema. Ulceration. Tendency to spontaneous bleeding.
Time Frame: 3 months
Population: Numbers indicate participants that were evaluable at 3 months.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Number analyzed (Participants) | 267 | 265
score on a scale | 0.141 (0.0046) | 0.154 (0.0046)

2. Primary Outcome: Change From Baseline in Löe-Silness Gingivitis Index
Description: as for outcome 1
Time Frame: 2 months
Population: Numbers indicate the participants that were evaluable at 2 months.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Number analyzed (Participants) | 278 | 270
score on a scale | 0.124 (0.0044) | 0.137 (0.0045)

3. Primary Outcome: Change From Baseline in Löe-Silness Gingivitis Index
Description: as for outcome 1
Time Frame: 1 month
Population: Numbers indicate the participants that were evaluable at 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Number analyzed (Participants) | 275 | 273
score on a scale | 0.112 (0.0045) | 0.125 (0.0045)

4. Secondary Outcome: Gestational Age (Weeks)
Description: log[42.9-gestational age]
Time Frame: At delivery
Population: This data includes the number of subjects who had evaluable data for the obstetric measure (Gestational Age) was 613. Possible reasons for data being declared as non-evaluable includes: being dropped from the study, failing to have enough product for the duration of pregnancy, missing multiple visits, or failing other protocol criteria.
Measure: Least Squares Mean (Standard Error); unit: log weeks
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Number analyzed (Participants) | 311 | 302
log weeks | 1.3988 (0.03394) | 1.3271 (0.03403)

5. Other Pre Specified Outcome: Neonate Birth Weight (Grams)
Time Frame: At delivery
Measure: Least Squares Mean (Standard Error); unit: grams
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Number analyzed (Participants) | 311 | 301
grams | 3095.97 (46.588) | 3167.80 (45.955)

6. Other Pre Specified Outcome: Preterm Birth (Gestational Age < 37 Weeks)
Time Frame: At delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
Number analyzed (Participants) | 311 | 302
Participants | 32 | 21

ADVERSE EVENTS:
Time Frame: Participants were enrolled 8-24 weeks into pregnancy until delivery
Arm/Group | Regular Oral Hygiene | Advanced Oral Hygiene Plus Counseling
All-Cause Mortality (participants affected / at risk) | 0/373 | 0/373
Serious Adverse Events (participants affected / at risk) | 79/373 | 75/373
Other Adverse Events (participants affected / at risk) | 353/373 | 329/373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Regular Oral Hygiene (N=373) | Advanced Oral Hygiene Plus Counseling (N=373)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
CARDIOMEGALY (Cardiac disorders) | 1 | 0
FOETAL HEART RATE DECELERATION (Cardiac disorders) | 1 | 0
PULMONARY VALVE STENOSIS (Cardiac disorders) | 1 | 0
CHROMOSOMAL DELETION (Congenital, familial and genetic disorders) | 0 | 1
FALLOT'S TETRALOGY (Congenital, familial and genetic disorders) | 0 | 1
POLYDACTYLY (Congenital, familial and genetic disorders) | 1 | 1
PULMONARY ARTERY STENOSIS CONGENITAL (Congenital, familial and genetic disorders) | 0 | 1
RENAL APLASIA (Congenital, familial and genetic disorders) | 1 | 0
SICKLE CELL ANAEMIA WITH CRISIS (Congenital, familial and genetic disorders) | 0 | 1
TRANSPOSITION OF THE GREAT VESSELS (Congenital, familial and genetic disorders) | 0 | 1
TRISOMY 21 (Congenital, familial and genetic disorders) | 2 | 0
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 1
NAUSEA (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 2
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 2
ALLOIMMUNISATION (Immune system disorders) | 0 | 1
RHESUS INCOMPATIBILITY (Immune system disorders) | 0 | 1
APPENDICITIS (Infections and infestations) | 1 | 0
CHORIOAMNIONITIS (Infections and infestations) | 14 | 10
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 1
MENINGITIS VIRAL (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 2
PYELONEPHRITIS (Infections and infestations) | 0 | 1
ABDOMINAL INJURY (Injury, poisoning and procedural complications) | 1 | 1
INTENTIONAL OVERDOSE (Injury, poisoning and procedural complications) | 0 | 1
BLOOD PRESSURE INCREASED (Investigations) | 3 | 1
CARDIAC MURMUR (Investigations) | 0 | 1
FOETAL HEART RATE ABNORMAL (Investigations) | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
FINGER DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
NOSE DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 1 | 0
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 0 | 1
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 2 | 3
ABORTION THREATENED (Pregnancy, puerperium and perinatal conditions) | 0 | 1
CERVICAL INCOMPETENCE (Pregnancy, puerperium and perinatal conditions) | 1 | 1
FOETAL DISTRESS SYNDROME (Pregnancy, puerperium and perinatal conditions) | 1 | 0
FOETAL GROWTH RESTRICTION (Pregnancy, puerperium and perinatal conditions) | 1 | 7
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 1 | 0
GESTATIONAL HYPERTENSION (Pregnancy, puerperium and perinatal conditions) | 8 | 7
HAEMORRHAGE IN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 0
HELLP SYNDROME (Pregnancy, puerperium and perinatal conditions) | 3 | 0
IMMINENT ABORTION (Pregnancy, puerperium and perinatal conditions) | 1 | 2
OLIGOHYDRAMNIOS (Pregnancy, puerperium and perinatal conditions) | 2 | 3
PLACENTA PRAEVIA HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 1 | 0
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 21 | 12
PREMATURE DELIVERY (Pregnancy, puerperium and perinatal conditions) | 27 | 15
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 6 | 7
PREMATURE RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 9 | 7
PREMATURE SEPARATION OF PLACENTA (Pregnancy, puerperium and perinatal conditions) | 2 | 1
STILLBIRTH (Pregnancy, puerperium and perinatal conditions) | 4 | 3
UTERINE CONTRACTIONS DURING PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 1 | 1
KETONURIA (Renal and urinary disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 0
PYELOCALIECTASIS (Renal and urinary disorders) | 0 | 2
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 4 | 3
ACUTE CHEST SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ABORTION INDUCED (Surgical and medical procedures) | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1
HYPERTENSION (Vascular disorders) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regular Oral Hygiene (N=373) | Advanced Oral Hygiene Plus Counseling (N=373)
ANAEMIA (Blood and lymphatic system disorders) | 35 | 41
NAUSEA (Gastrointestinal disorders) | 18 | 19
VOMITING (Gastrointestinal disorders) | 14 | 19
CHORIOAMNIONITIS (Infections and infestations) | 24 | 22
URINARY TRACT INFECTION (Infections and infestations) | 27 | 18
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 21 | 24
STREPTOCOCCUS TEST POSITIVE (Investigations) | 88 | 94
HEADACHE (Nervous system disorders) | 19 | 13
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 25 | 17
GESTATIONAL HYPERTENSION (Pregnancy, puerperium and perinatal conditions) | 19 | 19
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 23 | 15
PREMATURE DELIVERY (Pregnancy, puerperium and perinatal conditions) | 40 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Joint agreement with PIs.

DOCUMENTS (2):
  • Study Protocol (2013-04-08): https://cdn.clinicaltrials.gov/large-docs/87/NCT01549587/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT01549587/SAP_001.pdf